CLINICAL TRIAL: NCT02655848
Title: Long Head Biceps Tenodesis or Tenotomy in Arthroscopic Rotator Cuff Repair: An International Multicenter Prospective Randomized Clinical Trial
Brief Title: Tenotomy or Tenodesis of Long Head Biceps in Arthroscopic Rotator Cuff Repair
Acronym: BITE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Onze Lieve Vrouwe Gasthuis (Other)
Collaborators: Nederlandse Vereniging voor Arthroscopie (Unknown); Smith & Nephew, Inc. (Industry)
Responsible Party: Principal Investigator, DFP van Deurzen, Orthopedic Surgeon, Onze Lieve Vrouwe Gasthuis
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: WO 10.087
Record Dates: First submitted 2015-12-29; First posted 2016-01-14 (Estimated); Last update posted 2019-10-01 (Actual); Status verified 2019-09

CONDITIONS: Rotator Cuff Syndrome
Keywords: Popeye; Long Head Biceps Tendon; Arthroscopy; Functional result

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- @ Cuff repair with LHB tenodesis (Active Comparator): In case of pathologic changes of the long Head Biceps tendon, a tenodesis is performed in adjunct to performing an arthroscopic rotator cuff repair.
  Interventions: Procedure: Arthroscopic rotator cuff repair; Procedure: LHB Tenodesis
- @ cuff repair with LHB tenotomy (Active Comparator): In case of pathologic changes of the long Head Biceps tendon, a tenotomy is performed in adjunct to performing an arthroscopic rotator cuff repair.
  Interventions: Procedure: Arthroscopic rotator cuff repair; Procedure: LHB Tenotomy

INTERVENTIONS:
Procedure: Arthroscopic rotator cuff repair — Arthroscopic rotator cuff repair using suture anchors
Procedure: LHB Tenodesis — Arthroscopic tenotomy and subsequent fixation of long head biceps proximal in the biceps groove
  Arms: @ Cuff repair with LHB tenodesis
Procedure: LHB Tenotomy — Arthroscopic tenotomy of long head biceps
  Arms: @ cuff repair with LHB tenotomy

SUMMARY:
During arthroscopic rotator cuff (infraspinatus/supraspinatus) repair, biceps tendon lesions are frequently encountered. However, the most optimal treatment of the diseased long head of the biceps (LHB) tendon during rotator cuff repair remains a topic of debate: tenotomy or tenodesis. The hypothesis is that there is no difference in functional outcome between LHB tenotomy and LHB tenodesis when performed in adjunct to arthroscopic rotator cuff repair.

DETAILED DESCRIPTION:
Patients older than 50 years with a supraspinatus and/or infraspinatus tendon rupture sized smaller than 3cm, who are encountered with LHB pathology, will be randomized to either LHB tenotomy or LHB tenodesis. Clinical and self-reported data will be collected pre-operatively, and 6 weeks, 3 months, and 1 year after surgery.

Primary outcome is overall shoulder function evaluated with the Constant score. As additional measures of shoulder function, the Dutch Oxford Shoulder Test and the Disabilities of the Arm Shoulder and Hand questionnaire will be assessed. Other evaluations include cosmetic appearance evaluated by the ''Popeye'' deformity, arm cramping pain, elbow flexion strength, MRI evaluation, quality of life, and cost of surgery. To detect non-inferiority with a one-sided, two-sample t-test with a 80% power and a significance level (alpha) of 0.025, the required sample size is 98 patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 50 years
* Degenerative rotator cuff lesion of supraspinatus/infraspinatus tendon, smaller than three centimeter.
* Patients need to be able to read and write in Dutch or English language in order to complete the questionnaires, and sign informed consent.

Exclusion Criteria:

* Acute, traumatic or partial thickness rotator cuff rupture, or in case a full thickness tear is larger than 3 cm measured using an arthroscopic ruler.
* Accompanying subscapularis tendon lesion
* Hour-glass deformation bicepstendon origin or in case of accompanying subscapularis tendon rupture.
* Osteoarthritis of the glenohumeral joint
* Acromion to humeral head distance measuring 6mm or smaller.
* Prior surgery to the involved shoulder
* Dementia or inability to complete questionnaires and assessments

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2012-07; Primary Completion 2019-09 (Actual); Study Completion 2019-09 (Actual)

PRIMARY OUTCOMES:
Shoulder function quantified with the Constant score (0-100) | 1 year
  Sum of the items below:
  ADL: Patient reported shoulder function during work (0-4), recreation/sports (0-4), and sleep (0-2).
  Pain: Patient reported pain in the shoulder (severe=0,moderate=5,mild=10,no pain=15).
  ROM: Anteflexion up to waist(2)/xiphoid process(4)/neck(6)/head(8)/above head(10) Elevation in degrees: 0-30(0)/31-60(2)/61-90(4)/91-120(6)/121-150(8)/151-180(10) Abduction in degrees: 0-30(0)/31-60(2)/61-90(4)/91-120(6)/121-150(8)/151-180(10) External rotation: impossible to reach head with hand(0)/hand behind head-elbow forward(2)/hand behind head-elbow backward(4)/hand on head-elbow forward(6)/hand on head-elbow backward(8)/full elevation hand from head(10) Internal rotation: dorsal part of the hand reaching lateral thigh(0)/buttock(2)/lumbo-sacral junction(4)/L3(6)/Th12(8)/between scapulae(10).
  Abduction force at 90 degrees in pounds (max. 25)

SECONDARY OUTCOMES:
Popeye phenomenon | 1 year
  Presence of a Popeye deformity in the upper arm (yes/no), as reported by the patient, the treating surgeon, and a blinded assessor.
Cosmetic appearance | 1 year
  Patients will assess cosmetic appearance on a VAS scale.
MRI-based location of the biceps tendon | 1 year
  MRI imaging at 1 year after surgery will be used to assess the location of the proximal biceps tendon. Absence of the biceps tendon in the bicipital groove confirms a successfully performed LHB tenotomy. Absence of the biceps tendon in the bicipital groove confirms failed LHB tendodesis. In addition, the rotator cuff is classified as fully healed, partially healed or recurrent rupture.
Self-reported shoulder function | 1 year
  Patients will complete two validated questionnaires: the Disabilities of Arm, Shoulder and Hand Questionnaire (DASH) and the Dutch Oxford Shoulder Test (DOST)
Pain | 1 year
  Patients will be asked to report if they have pain (yes/no), and to indicate the level of pain on a VAS scale. The VAS scores will be recorded separately for general pain and for pain in the bicipital groove.
Elbow flexion strength | 1 year
  A dynamometer will be used to assess elbow flexion strength with the lower arm in full supination. The Elbow Strength Index is calculated by dividing the strength in the affected side by the strength in the contralateral side.
Quality of life | 1 year
  Patients will complete the validated questionnaire 'EQ-5D', which covers 5 domains (mobility, personal care, daily activities, pain and mood), as well as a 100 point thermometer on general health.
Post-operative status of rotator cuff | 1 year
  Based on MRI imaging at 1 year after surgery, the rotator cuff is classified as fully healed, partially healed or recurrent rupture.
Duration of surgery | 1 year
  The duration of surgery will be calculated based on the start and end times of each surgery.
Complications | 1 year
  All complications and serious adverse events in the study population are recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Derek van Deurzen, MD, Principal Investigator — OLVG
Locations (10):
- Netherlands (10):
  - Slootervaart ziekenhuis, Amsterdam
  - Kliniek De Lairesse, Amsterdam
  - OLVG, Amsterdam
  - Gelre ziekenhuis, Apeldoorn
  - Amphia ziekenhuis, Breda
  - Groene Hart Ziekenhuis, Gouda
  - Tergooi Ziekenhuizen, Hilversum
  - Spaarne Ziekenhuis, Hoofddorp
  - St Antonius, Nieuwegein
  - Canisius Wilehelmina Zkh, Nijmegen

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gurnani N, van Deurzen DF, Janmaat VT, van den Bekerom MP. Tenotomy or tenodesis for pathology of the long head of the biceps brachii: a systematic review and meta-analysis. Knee Surg Sports Traumatol Arthrosc. 2016 Dec;24(12):3765-3771. doi: 10.1007/s00167-015-3640-6. Epub 2015 May 15. PMID 25975753
- [Background] Zhang Q, Zhou J, Ge H, Cheng B. Tenotomy or tenodesis for long head biceps lesions in shoulders with reparable rotator cuff tears: a prospective randomised trial. Knee Surg Sports Traumatol Arthrosc. 2015 Feb;23(2):464-9. doi: 10.1007/s00167-013-2587-8. Epub 2013 Jul 5. PMID 23828089
- [Background] Galasso O, Gasparini G, De Benedetto M, Familiari F, Castricini R. Tenotomy versus tenodesis in the treatment of the long head of biceps brachii tendon lesions. BMC Musculoskelet Disord. 2012 Oct 22;13:205. doi: 10.1186/1471-2474-13-205. PMID 23088416
- [Derived] van Deurzen DF, Scholtes VA, Willigenburg NW, Gurnani N, Verweij LP, van den Bekerom MP; BITE collaboration group. Long head BIceps TEnodesis or tenotomy in arthroscopic rotator cuff repair: BITE study protocol. BMC Musculoskelet Disord. 2016 Aug 30;17(1):375. doi: 10.1186/s12891-016-1230-5. PMID 27577549